CLINICAL TRIAL: NCT02774330
Title: Impact of a Local Staple Foods Ordinance on Food Choice and Calories Purchased
Brief Title: Impact of the Minneapolis Staple Foods Ordinance
Acronym: STORE
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 1311S45924; 1410S54204 (Other: University of Minnesota Institutional Review Board); R01DK104348 (NIH); U48DP005022 (NIH)
Record Dates: First submitted 2016-05-04; First posted 2016-05-17 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Food Policy
MeSH Terms: interventions — Policy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minneapolis, Minnesota Customers: Minneapolis, Minnesota has a policy in place whereby minimum quantities and varieties of healthy food are required for all licensed food stores. The policy is our "intervention" condition.
  Interventions: Other: Policy
- St. Paul, Minnesota Customers: No policy exists in St. Paul, Minnesota. This is the control condition.

INTERVENTIONS:
Other: Policy — This local policy change (i.e., the Minneapolis Staple Foods Ordinance) establishes minimum stocking criteria for a wide array of healthy foods as a requirement of food store licensing. To our knowledge, it is the first and only policy of its kind in the U.S. This Staple Foods Ordinance requires stores to stock specific types of foods in minimum quantities and varieties, including fruits and vegetables, low-fat dairy, and whole grains. A full list of all requirements can be found online through the City of Minneapolis: http://www.minneapolismn.gov/health/living/eating/staple-foods.
  Groups: Minneapolis, Minnesota Customers

SUMMARY:
Improving healthy food availability and decreasing the availability of high calorie, low nutrient products, particularly in underserved communities, has been identified as a leading strategy for local governments to prevent obesity. However, policy action in this area to date has been limited. This R01 will examine the impact of a local policy change that establishes minimum stocking criteria for a wide array of healthy foods as a requirement of food store licensing. To our knowledge, this is the only policy of its kind in the US. As such, if it is successful, it could serve as an important model policy for other local governments seeking to increase healthy food availability and prevent obesity through local policy action.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of a local policy change (i.e., the Minneapolis Staple Foods Ordinance) that establishes minimum stocking criteria for a wide array of healthy foods as a requirement of food store licensing. Recent calls to action from the Institute of Medicine, the Centers for Disease Control and Prevention and other authorities have identified improving access to healthy foods as a primary strategy for local governments to use in advancing obesity prevention efforts, but policy initiatives in this area have been limited. In this study, the impact of the Minneapolis Staple Foods Ordinance will be evaluated by assessing objectively measured changes in: (a) food environments among small- to mid-sized, urban food stores, including availability, promotion, advertising, quality, price, and placement of both healthy and unhealthy foods and beverages, (b) nutritional quality of consumer purchases at small food stores, including assessment of energy density and calories via customer intercept surveys and direct observation of purchases and (c) home food environments, including availability of healthy and unhealthy foods/beverages and an overall home food obesogenicity score, among households that frequently shop at small- to mid-sized stores. These changes will be assessed pre-policy implementation, as well as 4-, 12- and 24-months post-policy implementation, in two Minnesota cities: Minneapolis and St. Paul, (our control community). The proposed scope of work in this study is important because its takes advantage of a unique opportunity to evaluate an innovative local policy addressing a recommended action area for obesity prevention that aligns with key recommendations by leading obesity prevention authorities. To our knowledge, the Minneapolis Staple Food Ordinance is the only policy of its kind in the US, and as such it could serve as an important model policy for other local governments if it is successful.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must be able to speak and understand English
* Must have purchased at least one food or beverage item from a randomly selected store that meets the following criteria:
* Outside the central downtown commercial core
* Not authorized to accept benefits from the Special Supplemental Nutrition Program for Women, Infants, and Children
* Valid licensing address
* >100 square feet of retail floor space
* Not small vendors in market areas or specialty stores
* Non-supermarket
* Permission from store staff to recruit participants

Exclusion Criteria:

* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Customers exiting small- to mid-size food stores after having purchased a food or beverage item
Sampling Method: Non-Probability Sample
Enrollment: 3488 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12-18 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Healthy Food Supply (store-level) | 24 months post-policy implementation (i.e., 12-months post-policy enforcement)
  To assess changes in healthy and unhealthy food availability, we will use a tool developed at the Yale Rudd Center for Food Policy and Obesity to evaluate the impact of 2009 Special Supplemental Nutrition Program for Women, Infants, and Children policy revisions in small stores, with minor adaptations to suit the needs of our study (See Andreyeva et al, J Acad Nutr Diet. 2012;112(6):850-858). As detailed in Andreyeva et al, we will create and use an an adapted Healthy Food Supply (HFS) score that summarizes availability, price, quality, and variety in the stores in our sample.We will examine changes in healthy food supply scores over time in stores in our sample in Minneapolis (where the policy is in place, i.e., our "intervention" community) versus those in St. Paul (where no such policy exists, i.e., our "control" community).
Calories purchased (customer-level) | 24 months post-policy implementation (i.e., 12-months post-policy enforcement)
  Our staff will examine all foods and beverages purchased (via a "bag check") by participating customers existing stores in our sample and will record item names, product types and weights/sizes. We will conduct detailed nutrient analyses on these purchases to assess total calories purchased and possible changes in calories purchased over time, comparing relative changes in purchasing among participants recruited outside of stores in Minneapolis (where the policy is in place, i.e., our "intervention" community) versus those in St. Paul (where no such policy exists, i.e., our "control" community).

OTHER OUTCOMES:
Healthy home food availability/obesogenicity score (customer-level) | 24 months post-policy implementation (i.e., 12-months post-policy enforcement)
  Trained staffers will visit the homes of participants who report frequently shopping in small- and non-traditional food stores to complete a home food inventory using a validated assessment tool. (See Fulkerson et al, International Journal of Behavioral Nutrition and Physical Activity 2008;5(55).) Data collected using this tool will be used to create a validated summative obesogenicity score, as detailed in Fulkerson et al 2008. Changes in this score will be examined over time.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa N Laska, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Division of Epidemiology and Community Health, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caspi CE, Winkler MR, Lenk KM, Harnack LJ, Erickson DJ, Laska MN. Store and neighborhood differences in retailer compliance with a local staple foods ordinance. BMC Public Health. 2020 Feb 4;20(1):172. doi: 10.1186/s12889-020-8174-2. PMID 32019508
- [Derived] Laska MN, Caspi CE, Lenk K, Moe SG, Pelletier JE, Harnack LJ, Erickson DJ. Evaluation of the first U.S. staple foods ordinance: impact on nutritional quality of food store offerings, customer purchases and home food environments. Int J Behav Nutr Phys Act. 2019 Sep 18;16(1):83. doi: 10.1186/s12966-019-0818-1. PMID 31533737
- [Derived] Caspi CE, Lenk K, Pelletier JE, Barnes TL, Harnack L, Erickson DJ, Laska MN. Association between store food environment and customer purchases in small grocery stores, gas-marts, pharmacies and dollar stores. Int J Behav Nutr Phys Act. 2017 Jun 5;14(1):76. doi: 10.1186/s12966-017-0531-x. PMID 28583131

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-31): https://cdn.clinicaltrials.gov/large-docs/30/NCT02774330/Prot_SAP_000.pdf